CLINICAL TRIAL: NCT05189574
Title: Endoscopic Negative Pressure Therapy for Post-sleeve Gastrectomy Proximal Staple Line Leaks
Brief Title: Endo-Vac-Therapy for Post-Sleeve Gastrectomy Leaks
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Markus Reiser, M.D., Chief Dept. Gastroenterology, Ruhr University of Bochum
Other Study IDs: EVac-LSGL
Record Dates: First submitted 2021-12-19; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Anastomotic Leak
Keywords: staple line leak; endoscopic vacuum therapy; endoscopic negative pressure therapy; laparoscopic sleeve gastrectomy
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic negative pressure therapy — Endoscopic placement of a sponge in/at staple line leaks under negative pressure.

SUMMARY:
Endoscopic negative pressure therapy (ENPT) is a safe technique, showing promising results in the treatment of leakages of the upper and lower gastrointestinal tract. The purpose of this study is to determine the safety and efficacy of ENPT in the management of proximal staple line leak after sleeve gastrectomy.

DETAILED DESCRIPTION:
Clinical data of 40 cases of post-SG proximal staple line leak treated with ENPT are analysed. Success is defined as resolution of the fistula with no further need for intervention (surgical or endoscopic).

ELIGIBILITY:
Inclusion Criteria:

* Staple line leak detected by endoscopy and/or CT within 30 days after surgery.
* Age 18 years or older.
* Written informed consent.

Exclusion Criteria:

* Declined informed consent.
* Leaks detected later than 30 days after surgery.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older 18 years who underwent laparoscopic sleeve gastrectomy for morbid obesity and developed a proximal staple line leak within 30 days.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Number of patients with closure of staple line leak | up to 16 weeks
  Resolution of the fistula with no further need for intervention (surgical or endoscopic).

SECONDARY OUTCOMES:
Number of endoscopic interventions | up to 16 weeks
  Number of endoscopic interventions in each patient
Hospital stay | up to 24 weeks
  Time of hospital stay for each patient
Mortality | up to 24 weeks
  Mortality rate during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Markus Reiser, MD, Principal Investigator — Chief Dept. Medicine and Gastroenterology
Locations (1):
- Klinikum Vest GmbH, Recklinghausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No